CLINICAL TRIAL: NCT00608842
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of ATX-101 (Sodium Deoxycholate for Injection) Intralipomal Injections for the Treatment of Superficial Lipomas
Brief Title: Phase 2 Study for the Treatment of Superficial Lipomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kythera Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATX-101-07-05
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-12

CONDITIONS: Lipoma
MeSH Terms: conditions — Lipoma | interventions — Deoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Deoxycholic Acid 1% (Experimental): Participants received 1.0% deoxycholic acid administered at a volume dependent on the size of the lipoma, up to a maximum of 4.8 mL per treatment session, at 28-day intervals for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic Acid Injection
- Deoxycholic Acid 2% (Experimental): Participants received 2.0% deoxycholic acid administered at a volume dependent on the size of the lipoma, up to a maximum of 4.8 mL per treatment session, at 28-day intervals for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic Acid Injection
- Deoxycholic Acid 4% (Experimental): Participants received 4.0% deoxycholic acid administered at a volume dependent on the size of the lipoma, up to a maximum of 4.8 mL per treatment session, at 28-day intervals for up to a maximum of 4 treatments.
  Interventions: Drug: Deoxycholic Acid Injection
- Placebo (Placebo Comparator): Participants received matching vehicle placebo administered at a volume dependent on the size of the lipoma, up to a maximum of 4.8 mL per treatment session, at 28-day intervals for up to a maximum of 4 treatments.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Deoxycholic Acid Injection — Administered via intralipomal injection.
  Other Names: sodium deoxycholate; ATX-101
  Arms: Deoxycholic Acid 1%; Deoxycholic Acid 2%; Deoxycholic Acid 4%
Drug: Placebo — Matching vehicle placebo administered via intralipomal injection.
  Arms: Placebo

SUMMARY:
The purpose of this research is to compare the safety and effectiveness of 3 different concentrations of deoxycholic acid for injection against a placebo in the treatment of superficial lipomas.

DETAILED DESCRIPTION:
A lipoma is a fatty lump typically located on the trunk, shoulder, arms, or legs. For the purposes of this study, only lipomas on the trunk, arms, legs, or neck were treated. (Lipomas on the face, wrists, hands, lower portion of the spine, genitals, ankles, or feet were not treated.)

ELIGIBILITY:
Inclusion Criteria:

* One or more lipomas, based on clinical and histological diagnosis, which are accessible for treatment and assessment, are quantifiable along at least 2 perpendicular diameters, and have the following characteristics:

  * History of slow growth followed by dormancy, and stable for at least 6 months
  * Greatest length multiplied by greatest perpendicular width between 1 and 16 cm², inclusive
  * Discrete, oval to rounded in shape, not hard or attached to underlying tissue
  * Without changes in overlying skin (ie, inflammation, pain or tenderness, hyperpigmentation)
  * Located on the trunk, arms, legs, or neck
* Signed informed consent.

Exclusion Criteria:

* Absence of significant medical conditions that could affect safety
* History of surgical or deoxycholate treatment for lipomas
* Treatment with an investigational agent within 30 days before ATX-101 treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2007-11; Primary Completion 2008-08 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia S. Walker, M.D., Ph.D., Study Director — Kythera Biopharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Gary D. Monheit, M.D., Birmingham, Alabama
  - Stacy R. Smith, San Diego, California
  - Steven Grekin, D.O., Warren, Michigan
  - Joel Schlessinger, M.D., Omaha, Nebraska
  - David J. Goldberg, M.D., Westwood, New Jersey
  - Neil S. Sadick, M.D., New York, New York
  - Michael H. Gold, M.D., Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received matching placebo administered at a volume dependent on the size of the lipoma, up to a maximum of 4.8 mL per treatment session, at 28-day intervals for up to a maximum of 4 treatments.
Period: Overall Study
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Started | 15 | 15 | 15 | 17
Completed | 14 | 14 | 13 | 16
Not Completed | 1 | 1 | 2 | 1
Not completed — Participant's Request | 0 | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (MITT) population included all randomized participants who had received at least 1 dose of study material and who had at least 1 postbaseline observation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 14 | 17 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (9.5) | 48.5 (9.1) | 49.5 (10.5) | 45.5 (8.9) | 47.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 3 | 6 | 19
  Male | 10 | 10 | 11 | 11 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Severity of AEs was determined using the following scale:
  Mild: The participant was aware of a sign or symptom, but it was easily tolerated; Moderate: Discomfort or interference with usual activity; Severe: Incapacitating, with inability to engage in usual activity. The investigator determined the relationship of each AE to the administration of study material by answering the question: "Was there a reasonable possibility that the event may have been caused by treatment with study material?" A serious AE was an event that constituted a significant medical hazard or side effect, regardless of the investigator's or sponsor's opinion regarding relatedness to study material. Serious AEs included any event that was fatal or life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or other significant medical hazard.
Time Frame: Up to 24 weeks
Population: Safety population (all participants who received at least 1 dose of study medication)
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 17
participants
  Any adverse event | 12 | 13 | 14 | 12
  Any treatment-related adverse event | 6 | 9 | 8 | 7
  Any serious adverse event | 1 | 0 | 1 | 0
  Any severe adverse event | 1 | 1 | 2 | 0
  Any adverse event leading to drug discontinuation | 1 | 0 | 3 | 0

2. Secondary Outcome: Percentage of Participants With Complete Clearance or ≥ 75% Clearance
Description: At randomization 1 to 3 lipomas were selected for treatment. Lipomas were measured in 3 dimensions (longest length, perpendicular width, and height if possible) using digital calipers.
  Complete clearance indicates target lipoma(s) not present or detectable, and ≥ 75% clearance is defined as a ≥ 75% reduction from baseline in the area of target lipoma(s).
  For participants with > 1 target lipoma, the total area of all target lipomas was used in the calculation of response.
Time Frame: Baseline and week 20 (8 weeks after last dose)
Population: MITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 17
percentage of participants
  Complete Clearance | 0.0 | 0.0 | 7.1 | 0.0
  ≥ 75% Cleared | 13.3 | 6.7 | 14.3 | 11.8
Statistical Analysis 1: Comparison: Deoxycholic Acid 1% vs Placebo; Complete Clearance; Test type: Superiority or Other; Difference to placebo = 0.0, 95% CI 2-sided [-18.4 to 20.4]
Statistical Analysis 2: Comparison: Deoxycholic Acid 2% vs Placebo; Complete Clearance; Test type: Superiority or Other; Difference to placebo = 0.0, 95% CI 2-sided [-18.4 to 20.4]
Statistical Analysis 3: Comparison: Deoxycholic Acid 4% vs Placebo; Complete Clearance; Test type: Superiority or Other; Difference to placebo = 7.1, 95% CI 2-sided [-12.2 to 31.5]
Statistical Analysis 4: Comparison: Deoxycholic Acid 1% vs Placebo; ≥ 75% Cleared; Test type: Superiority or Other; Difference to placebo = 1.6, 95% CI 2-sided [-23.0 to 27.5]
Statistical Analysis 5: Comparison: Deoxycholic Acid 2% vs Placebo; ≥ 75% Cleared; Test type: Superiority or Other; Difference to placebo = -5.1, 95% CI 2-sided [-28.3 to 19.6]
Statistical Analysis 6: Comparison: Deoxycholic Acid 4% vs Placebo; ≥ 75% Cleared; Test type: Superiority or Other; Difference to placebo = 2.5, 95% CI 2-sided [-22.3 to 29.5]

3. Primary Outcome: Number of Participants With Newly Occurring or Worsening Biochemistry/Hematology/Urinalysis Abnormalities
Description: An abnormality is defined as a value outside the limits of the expanded normal range/notable range.
Time Frame: 24 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 17
participants
  Blood triglycerides | 0 | 0 | 1 | 0
  Alanine transaminase | 0 | 0 | 1 | 0
  Aspartate aminotransferase | 0 | 0 | 1 | 0
  Alkaline phosphatase | 0 | 0 | 1 | 0
  Urinalysis - Glucose | 0 | 0 | 1 | 0

4. Secondary Outcome: Percent Change From Baseline in the Sum of the Areas of All Treated Lipomas
Description: Percent change from baseline was calculated as the baseline total lipoma area - postbaseline total lipoma area / baseline total lipoma area * 100. A positive change indicates a reduction in size.
Time Frame: Baseline and week 12 (last treatment session), week 16 (4 weeks after last treatment), and week 20 (8 weeks after last treatment)
Population: MITT Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Number analyzed (Participants) | 15 | 15 | 14 | 17
percent change
  Week 12 | 41.2 (31.5) | 28.5 (46.0) | 18.0 (34.9) | 38.5 (32.4)
  Week 16 | 43.9 (30.1) | 23.3 (41.8) | 20.0 (38.2) | 32.1 (40.5)
  Week 20 | 50.1 (30.6) | 25.9 (42.6) | 35.9 (40.7) | 36.7 (38.0)

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs or Weight
Time Frame: Up to 24 weeks
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 17
participants | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Positive Histopathology Results at Screening
Description: A needle core tissue sample biopsy was performed at screening for all treated lipomas.
Time Frame: Screening (prior to randomization)
Population: Safety population with biopsy results at screening
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Number analyzed (Participants) | 13 | 12 | 13 | 14
participants
  Acute inflammation | 0 | 0 | 1 | 0
  Chronic inflammation | 0 | 0 | 0 | 0
  Fibrosis/scarring | 0 | 0 | 1 | 0
  Hemorrhage | 0 | 0 | 2 | 1
  Mature adipose tissue | 11 | 11 | 13 | 13
  Necrosis | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Positive Histopathology Results at Week 20
Description: After the completion of all tests and procedures scheduled for week 20, participants with treated lipomas that remained palpable could have their treated lipomas excised.
Time Frame: Week 20
Population: Safety population with biopsy results at week 20
Measure: Number; unit: participants
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Number analyzed (Participants) | 15 | 13 | 15 | 16
participants
  Acute inflammation | 3 | 2 | 1 | 0
  Chronic inflammation | 10 | 12 | 13 | 0
  Fibrosis/scarring | 13 | 12 | 14 | 6
  Hemorrhage | 5 | 5 | 6 | 2
  Mature adipose tissue | 15 | 13 | 15 | 16
  Necrosis | 14 | 13 | 14 | 3

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Deoxycholic Acid 1% | Deoxycholic Acid 2% | Deoxycholic Acid 4% | Placebo
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 1/15 | 0/17
Other Adverse Events (participants affected / at risk) | 12/15 | 13/15 | 14/15 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid 1% (N=15) | Deoxycholic Acid 2% (N=15) | Deoxycholic Acid 4% (N=15) | Placebo (N=17)
Patella Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tibia Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Breast Cancer (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deoxycholic Acid 1% (N=15) | Deoxycholic Acid 2% (N=15) | Deoxycholic Acid 4% (N=15) | Placebo (N=17)
Injection Site Erythema (General disorders) | 6 | 6 | 4 | 3
Injection Site Bruising (General disorders) | 3 | 4 | 6 | 5
Injection Site Pain (General disorders) | 3 | 4 | 5 | 3
Injection Site Induration (General disorders) | 2 | 3 | 3 | 3
Injection Site Anaesthesia (General disorders) | 2 | 3 | 2 | 3
Injection Site Discolouration (General disorders) | 3 | 3 | 3 | 1
Injection Site Pruritus (General disorders) | 3 | 3 | 1 | 0
Injection Site Swelling (General disorders) | 2 | 1 | 3 | 1
Injection Site Irritation (General disorders) | 1 | 1 | 2 | 1
Injection Site Ulcer (General disorders) | 2 | 0 | 2 | 0
Injection Site Discharge (General disorders) | 1 | 1 | 1 | 0
Injection Site Haemorrhage (General disorders) | 2 | 0 | 0 | 1
Injection Site Desquamation (General disorders) | 1 | 0 | 0 | 0
Injection Site Inflammation (General disorders) | 1 | 0 | 0 | 0
Injection Site Rash (General disorders) | 1 | 0 | 0 | 0
Injection Site Warmth (General disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 3 | 3 | 2
Influenza (Infections and infestations) | 3 | 0 | 1 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 2
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Tinea Infection (Infections and infestations) | 0 | 0 | 0 | 1
Vaginitis Bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle Strain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Jaundice (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Infection (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood Cholesterol Increased (Investigations) | 0 | 0 | 0 | 1
Blood Triglycerides Increased (Investigations) | 0 | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1 | 0
Urine Colour Abnormal (Investigations) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Hepatitis C (Hepatobiliary disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical study agreement requires that the investigator or institution obtain written consent from Kythera Biopharmaceuticals, Inc. prior to presenting and/or publishing results of this study.